CLINICAL TRIAL: NCT03655067
Title: Use of an Internet-Based Cognitive Behavioral Therapy Intervention (CATCH-IT) for the Treatment of Depressive Symptoms in Adolescents With Type 1 Diabetes Mellitus
Brief Title: Internet-Based Cognitive Behavioral Therapy for Depressive Symptoms in Adolescents With Type 1 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Ellen Grishman, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU-2020-0230
Record Dates: First submitted 2018-08-21; First posted 2018-08-31 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Type 1 Diabetes Mellitus; Depressive Symptoms
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Depression

STUDY DESIGN:
Intervention Model Description: Participants will be randomized at the baseline visit to the CATCH-IT Intervention or Control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The participants in the Intervention group will receive the CATCH-IT program which consists of a motivational component and the internet program for the adolescent. The participants in the Intervention group will receive motivational interviewing at their baseline visit as well as motivational coaching with safety phone calls during weeks 1-6.
  Interventions: Behavioral: CATCH-IT
- Usual Care (No Intervention): Participants in the Usual Care group may undergo an evaluation with the Social Worker if the clinician determines that it is necessary. The participants in the Usual Care group will also receive motivational coaching with safety phone calls during weeks 1-6.

INTERVENTIONS:
Behavioral: CATCH-IT — The CATCH-IT internet program consists of 14 modules and exercises and activities based on best practices components of depression prevention. They will be instructed to complete at least 2 modules a week, over a period of 6 weeks. This would require at least 40 minutes per week (approximately 20 minutes minimum per module).
  Arms: Intervention

SUMMARY:
This study evaluates the use of an established internet-based cognitive behavioral therapy intervention in a group of adolescents with type 1 diabetes and mild to moderate depressive symptoms. Half of the participants will receive the internet-based intervention while the other half will receive usual care.

DETAILED DESCRIPTION:
Adolescents with diabetes have a higher incidence of subclinical and clinical depression compared to healthy adolescents. Patients with diabetes who are clinically or subclinically depressed are at high risk for poor glycemic control.

Studies evaluating prevention and treatment strategies for depression in patients with type 1 diabetes have shown that group cognitive-behavioral therapy (CBT) and individual interpersonal psychotherapy (IPT) can reduce the risk of depressive illness in adolescents with diabetes. Computerized interventions show evidence of being efficacious, and have been recommended as the "first line" intervention.

The Competent Adulthood Transition with Cognitive Humanistic and Interpersonal Teaching (CATCH-IT) internet program has shown positive results with adolescents at risk for depression, but has not been used in patients with a chronic illness like diabetes. CATCH-IT is based on established CBT and IPT treatment models. It includes a) an innovative and effective brief practitioner-provided motivation enhancement component (in person at enrollment and through phone calls) and b) self-directed modules for the adolescent that can be accessed on the internet.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-17 receiving ongoing medical care in the Diabetes Clinic at Children's Medical Center Dallas.
* Patients must be fluent in English (the materials on the site have not been validated in any other language), be in at least the 8th grade, report/demonstrate comfort with use of a computer, and regular, convenient and discreet access to the internet.
* Patients must experience at least sub-threshold depression (CES-D score > 15).
* Patients must have had the diagnosis of type 1 diabetes for at least 12 months.

Exclusion Criteria:

* Patients who are medically unstable during their diabetes clinic visit will be excluded (i.e. diabetes ketoacidosis, symptomatic hypoglycemia).
* Patients who are too severely depressed for this form of intervention (i.e. meet criteria for MDD, endorse suicidal intent, PHQ-A score ≥ 20), those with a diagnosis or symptoms of severe mental illness (schizophrenia, bipolar disorder), prior psychiatric hospitalization, prior self-harm attempt.
* Patients receiving ongoing counseling or therapy services within the last year, by a licensed professional (counselor, psychologist or psychiatrist).
* Patients who are currently taking or begin taking psychotropic medications during study participation will be excluded/withdrawn.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Center for Epidemiological Studies - Depression Scale (CES-D) | 6 weeks
  A screening test for depression and depressive disorder. The CESD measures symptoms defined by the American Psychiatric Association' Diagnostic and Statistical Manual (DSM-V) for a major depressive episode.

SECONDARY OUTCOMES:
Hemoglobin A1c | 12 weeks
  Hemoglobin A1c- a 3-month surrogate marker of diabetes control
Patient Health Questionnaire Modified for Teens | 6 weeks and 12 weeks
  A self-completion screening questionnaire designed to detect symptoms of depression and suicide risk in adolescents.
Problem Areas in Diabetes - Teen version | 6 weeks and 12 weeks
  A validated measure of diabetes distress designed specifically for adolescents with type 1 diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Olga T Gupta, MD, Principal Investigator — UTSW
Locations (1):
- Children's Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No